CLINICAL TRIAL: NCT06226688
Title: Biofeedback Training on Shoulder Muscles Strength Post Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Ahmed Mahmoud Souliman, Demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004823; 202309250044 (Registry Identifier: Baheya research center)
Record Dates: First submitted 2024-01-14; First posted 2024-01-26 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: RCT 2 groups One of them control group And the other is study group
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Affected arm at the same side of mastectomy (Experimental): There is 2 arms Arm1:-arm at side of mastectomy without lymphedema trained by biofeedback
  Interventions: Procedure: Biofeedback device and other group control group; Procedure: Control group
- 2 arms one trained by biofeedback and other control without biofeedback (Experimental): Arm2:-arm at side of mastectomy on other group but not trained with biofeedback Training using shoulder ladder ,shoulder wheel ,shoulder mobilization and IPC
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Biofeedback device and other group control group — Intervention 1 :-Using the biofeedback device with dumble to strength affected arm post mastectomy
  Other Names: Expirmental trial by biofeedback device
  Arms: Affected arm at the same side of mastectomy
Procedure: Control group — Shoulder mobilization Shoulder ladder ex Shoulder wheel ex Ipc
  Other Names: Intervention 2 :- using traditional PT programme without using biofeedback

SUMMARY:
PURPOSE:The purpose of the study is to evaluate the effect of biofeedback on shoulder muscles strength post mastectomy.

BACKGROUND:

* The most common complications following mastectomy are pain, ipsilateral lymphedema of the upper limb (UL), reduced range of motion (ROM) of the shoulder, flexion and abduction is limited to 90°, and external rotation is limited to 40°, and there are postural changes
* One of the most common complications after breast cancer surgery is a functional limitation of the upper body. Up to 67% of breast cancer patients experience arm or shoulder impairment, including pain, numbness, loss of strength, and reduced ROM, after surgery
* Shoulder problems in breast cancer patients affect their daily activities, such as pulling a sweater overhead, fastening a bra, zipping up a back zipper, reaching overhead, and carrying heavy bags.
* Biofeedback is a mind-body technique in which individuals learn how to modify their physiology for the purpose of improving physical, mental, emotional and spiritual health. Much like physical therapy, biofeedback training requires active participation on the part of patients and often regular practice between training sessions. Clinical biofeedback may be used to manage disease symptoms as well as to improve overall health and wellness through stress management training. Research has shown that biofeedback interventions are efficacious in treating a variety of medical conditions, and many Americans are turning to biofeedback and other less traditional therapies for their (Dana et al., 2010).

HYPOTHESES: null hypothesis

RESEARCH QUESTION: Does biofeedback give effect on shoulder muscles strength post mastectomy?

DETAILED DESCRIPTION:
27 patient per group to G power 90% a Inclusion Criteria:

The subject selection will be according to the following criteria:

* Female patients with age range between 40-60 will participate in the study.
* All patients with their informed consent.
* All patients with unilateral mastectomy
* All patients have shoulder muscle weakness within 2 to 4 months post mastectomy
* All patients with chemo or radio therapy 1.2.b Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

* metastasis
* Psychological Disorder
* Lymphedema
* Neurological or musculoskeletal disorders

ELIGIBILITY:
Inclusion Criteria:

* The subject selection will be according to the following criteria:
* Female patients with age range between 40-60 will participate in the study.
* All patients with their informed consent.
* All patients with unilateral mastectomy
* All patients have shoulder muscle weakness within 2 to 4 months post mastectomy
* All patients with chemo or radio therapy

Exclusion Criteria:

* The potential participants will be excluded if they meet one of the following criteria:
* metastasis
* Psychological Disorder
* Lymphedema
* Neurological or musculoskeletal disorders

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Measure before and after shoulder muscles strength by hand held dynamometer | 6 wweks
  Measuring

CONTACTS AND LOCATIONS:
Overall Officials: Research ethical commity Physical therapy Cairo university, Principal Investigator — Research ethical commity
Locations (2):
- Egypt (2):
  - Nourhan Souliman, Cairo, Bahyea Foundation For Breast Cancer
  - Nourhan Ahmed mahmoud souliman, Cairo